CLINICAL TRIAL: NCT07168421
Title: LANdiolol to Avoid TAchycardia in Patients at Risk for Cardiovascular Events Undergoing Major Non-cardiac Surgery: a Feasibility Trial
Brief Title: LANdiolol to Avoid TAchycardia in Patients at Risk for Cardiovascular Events Undergoing Major Non-cardiac Surgery
Acronym: LANTA-P
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BECD-1-21
Record Dates: First submitted 2025-08-11; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Perioperative Myocardial Injury; Autonomic Dysfunction; Cardiovascular (CV) Risk; Major Surgery; Beta Blocker; Myocardial Injury After Non-cardiac Surgery
Keywords: perioperative myocardial injury; major surgery; beta blocker; myocardial injury after non-cardiac surgery; autonomic dysfunction
MeSH Terms: conditions — Primary Dysautonomias | interventions — landiolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Landiolol (Experimental): Landiolol will be titrated to keep heart rate below 90 beats per minute during surgery after exclusion of other factors possibly causing tachycardia (such as hypovolaemia or pain). Mean arterial pressure will be kept above 65 millimeters of mercury.
  Interventions: Drug: Landiolol
- Usual care (No Intervention): In the usual care group, mean arterial pressure will be maintained above 65 millimeters of mercury. In case of tachycardia, causing reasons (such as hypovolaemia) will be sought and treated.

INTERVENTIONS:
Drug: Landiolol — The main dose range is 1-40 mcg/kg/min, titrated to the effect on heart rate aiming for a heart rate of below 90 beats per minute throughout. This dose can be decreased to 0 if heart rate stays below target.
  Arms: Landiolol

SUMMARY:
Limiting perioperative tachycardia (aiming for a heart rate <90 beats per minute throughout the perioperative period) using the ultra-short acting beta-blocker landiolol in patients with cardiovascular risk factors undergoing major surgery might lower the incidence of perioperative myocardial injury. Feasibility of the intervention needs to be proven prior to conduction of a larger trial.

DETAILED DESCRIPTION:
Despite advances in surgical and anaesthetic techniques, perioperative mortality remains high, even in developed countries. Major complications contributing almost half of all deaths after surgery are major bleeding (17%), myocardial injury after non-cardiac surgery (13%) and sepsis (12%). Myocardial injury after non-cardiac surgery occurs up to 18% in patients >45 years and is associated with a marked increase in 30-day mortality. Additional factors posing patients at risk for perioperative myocardial injury might be autonomic dysfunction, measured as exaggerated heart rate response to exercise or impaired heart rate recovery thereafter, as perioperative tachycardia is associated with perioperative myocaridal injury. The perioperative use of beta-blockers remains controversial, but the newely marketed ultra-short acting and highly cardioselective beta-blocker landiolol offers the opportunity to reduce perioperative heart rate without affecting blood pressure. The intervention (perioperative reduction of heart rate using landiolol) in this specific patient population needs to be proven as feasible prior to conducting a larger scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective non-cardiac surgery defined as intermediate or high-risk by the 2022 european society of cardiology (ESC) guidelines
* expected duration of surgery of at least 90 minutes;
* expected length of hospital stay ≥ 24 hours;
* age > 45 years with at least two of the following risk factors (adapted from revised cardiac risk index):

  * ischemic heart disease (history of myocardial infarction or positive exercise test, current complaint of chest pain considered to be secondary to myocardial ischemia, use of nitrates, pathological Q waves, prior coronary revascularization);
  * history of congestive heart failure;
  * history of cerebrovascular disease;
  * insulin-dependent diabetes mellitus;
  * creatinine > 176.8 mmol/l;
  * pre-operative NTproBNP > 200 pg/ml;
* excessive sympathetic outflow as proven by exercise testing:

  * impaired HR recovery (≤ 12 bpm within 1 minute after cessation of exercise); OR
  * exaggerated HR response (≥ 12 bpm after 1 minute of unloaded pedalling);

Exclusion Criteria:

* unable to consent or follow study procedures;
* absolute contraindications for exercise testing;
* pregnancy or intention to become pregnant;
* active cardiac conditions (such as unstable coronary syndromes, decompensated heart failure, significant arrhythmias, severe valvular disease);
* urgent / emergency surgery;
* already on β-blocker (within the last 30 days prior to recruitment);
* contraindication for β-blocker therapy (bradycardia (HR < 55 bpm), hypotension (systolic blood pressure < 100 mmHg), severe peripheral vascular disease, severe asthma, allergy, higher-degree atrioventricular block);
* severe preoperative anaemia (haemoglobin < 100 g/L) unless there is a plan set up and followed for correction prior to surgery;
* planned intermediate care or intensive care admission;
* prior enrolment in this trial.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Time perioperative heart rate in target range | From induction of anaesthesia until discharge from postanaesthetic care unit [percent of time heart rate within target range (<90 beats per minute)]
  As a marker of successful intervention, time perioperative heart rate in target range (below 90 beats per minute) will serve as primary outcome. The intervention is considered feasible if the heart rate stays at least 90% of the time within the target range during the perioperative period.

SECONDARY OUTCOMES:
Perioperative heart rate | From induction of anaesthesa until discharge from postanaesthetic care unit [heart rate in beats per minute * minutes ]
  Perioprative heart rate will be calculated as time weighted area under the curve for the perioperative period.
Dose of vasopressors | Induction of anaesthesia until discharge from postanaeshetic care unit [mcg per recorded drug]
  Total dose of vasopressors such as noradrenalin, ephedrine or phenylephrine will be recorded in micrograms.
Length of postanaesthetic care unit stay | Admission to postanaesthetic care unit until discharge from postanaesthetic care unit [minutes]
  Lenght of postaenaesthetic care unit stay will be recorded in minutes.
Length of hospital stay | Admission to hospital until discharge from hospital [days]
  Length of hospital stay will be recorded in days.
Perioperative myocardial injury | 72 hours after surgery
  Perioperative myocardial injury (PMI) is defined as an increase of hsTroponinT ≥ 14ng/L above the preoperative value according to the Basel-PMI criteria, not meeting major adverse cardiovascular event (MACE) criteria.

OTHER OUTCOMES:
Major adverse cardio- and cerebrovascular events | 30 days after surgery
  Major adverse cardio- and cerebrovascular events (MACCE) include diagnosis of non-fatal cardiac arrest, acute myocardial infarction, congestive heart failure, new cardiac arrhythmia or angina, non-fatal stroke.
All-cause death | 30 days after surgery
  This parameter serves to assess postoperative mortality.
Quality of life (EQ-5D) | 30 days after surgery
  Quality of life will be assessed using the EQ-5D questionnaire. The EQ-5D questionnaire is a standardised health-related quality of life questionnaire developed by the EuroQol Group. It assesses five dimensions of health and results in an utility index score ranging from 0 (death) to 1 (perfect health).
Comprehensive complication index | 30 days after surgery
  The comprehensive complication index is calculated as a sum of all complications weighted for their severity. It results in a continuous scale ranking the severity of any combination of complications from 0 (no complication) to 100 (death).

CONTACTS AND LOCATIONS:
Locations (1):
- Bern University Hospital, Freiburgstrasse, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
IPD can be provided on reasonable request